CLINICAL TRIAL: NCT04006470
Title: Bioavailable Stannous Fluoride Dentifrice Meta-Analyses: Effects on Dentine Hypersensitivity and Enamel Erosion
Brief Title: Meta-analysis of Stannous Fluoride and the Effects on Enamel Erosion
Status: Completed | Type: Observational
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019SnF2ErosionAnalysis
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Enamel Erosion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stannous Fluoride Dentifrice: Twice daily use
  Interventions: Drug: Stannous fluoride dentifrice
- Positive control dentifrice: Twice daily use
  Interventions: Drug: Positive control dentifrice
- Negative control dentifrice: Twice daily use
  Interventions: Drug: Negative control dentifrice

INTERVENTIONS:
Drug: Stannous fluoride dentifrice — Stannous fluoride (0.454%) dentifrice
  Groups: Stannous Fluoride Dentifrice
Drug: Positive control dentifrice — Positive control dentifrice containing potassium nitrate or arginine.
  Groups: Positive control dentifrice
Drug: Negative control dentifrice — Negative control dentifrice containing either sodium fluoride (0.243%) or sodium monofluorophosphate (0.76%)
  Groups: Negative control dentifrice

SUMMARY:
The aim of this 5 study analysis was to compare the effect of bioavailable stannous fluoride (SnF2) dentifrices to assess enamel erosion protection in-situ using surface profilometry.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This meta-analysis includes healthy adult male and females.
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Surface profilometry | 10 days
  Enamel samples will be measured via profilometry after 10 days of study use.

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple P&G Investigation Clinical Sites, Cincinnati, Ohio, United States